CLINICAL TRIAL: NCT02777567
Title: Open Label, Multicenter, Real World Treatment Study of Single Agent Tagrisso for Patients With Advanced/Metastatic Epidermal Growth Factor Receptor (EGFR) T790M Mutation-Positive Non-Small Cell Lung Cancer (NSCLC), Who Have Progressed on or After EGFR Tyrosine Kinase Receptor (TKI) Therapy
Brief Title: KOREA Study (Korea Osimertinib Real World Evidence Study to Assess Safety and Efficacy)
Acronym: KOREA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160R00009
Record Dates: First submitted 2016-05-13; First posted 2016-05-19 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of this study are to assess the safety and efficacy of single agent Tagrisso (Osimertinib, hereinafter "the study drug") in a real world setting in adult patients with advanced or metastatic, epidermal growth factor receptor (EGFR) T790M mutation-positive Non-Small Cell Lung Cancer (NSCLC), Who Have Progressed on or after EGFR tyrosine kinase receptor (TKI) therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Eligible for, or on active study drug treatment according to the approved label; patients with locally advanced or metastatic, EGFR T790M mutation-positive NSCLC, who have progressed on or after EGFR tyrosine kinase receptor (TKI) therapy
* 2. Provision of signed and dated written informed consent by the patient or legally acceptable representative

Exclusion Criteria:

* 1. History of hypersensitivity to excipients of the study drug or to drugs with a similar chemical structure or class to the study drug
* 2. Pregnancy and/or breast feeding
* 3. Current participation in any interventional trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with locally advanced or metastatic, EGFR T790M mutation-positive NSCLC, who have progressed on or after EGFR tyrosine kinase receptor (TKI) therapy
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Proportion (%) of patients with adverse events (AEs), serious adverse events (SAEs) and AEs of special interest (AESI) | up to one year
  Proportion (%) of patients with adverse events (AEs), serious adverse events (SAEs) and AEs of special interest (AESI)
Severity of (S)AEs | up to one year
  Severity of (S)AEs

SECONDARY OUTCOMES:
ORR (Objective response rate), if available | up to one year
  ORR (Objective response rate), if available
PFS (Progression free survival), if available | up to one year
  PFS (Progression free survival), if available

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, South Korea, South Korea, South Korea

REFERENCES:
- See also: redacted synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160R00009&attachmentIdentifier=92919e00-80b9-49a7-b77f-ff6dbe6d9738&fileName=D5160R00009_synopsis.pdf&versionIdentifier=